CLINICAL TRIAL: NCT06629012
Title: Breast Neurotization During Breast Reconstruction Enhances Quality of Life
Brief Title: Autologous Nerve Graft Breast Reconstruction Neurotization
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Professor, Chang Gung Memorial Hospital
Other Study IDs: 202101923B0-N
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Breast Reconstruction; Breast Cancer Patients; Nipple-sparing Mastectomy
Keywords: breast reconstruction; nipple-sparing mastectomy; breast neurotization; quality of life; autologous nerve graft; nipple sensation
MeSH Terms: interventions — Mammaplasty; Nerve Transfer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Innervated group: Patients received breast neurotization
  Interventions: Procedure: Breast reconstruction with neurotization
- Non-innervated group: Patients did not receive breast neurotization
  Interventions: Procedure: Breast reconstruction without neurotization

INTERVENTIONS:
Procedure: Breast reconstruction with neurotization — Patients received breast reconstruction with neurotization procedure
  Groups: Innervated group
Procedure: Breast reconstruction without neurotization — Patients received breast reconstruction without neurotization
  Groups: Non-innervated group

SUMMARY:
The goal of this observational study is to learn about the improvement of quality of life in accordance with breast neurotization in breast cancer patients. The patient-reported outcome was assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient who receive breast reconstruction
* Patient who is willing to fill in the questionnaire

Exclusion Criteria:

* Patient who receive breast reconstruction for the reason other than breast cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing nipple-sparing mastectomy and immediate breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-operative Quality of life | Before breast reconstructive surgery
  Patient-reported outcome assessed by the BREAST-Q™ Reconstruction module questionnaire and a additional questionnaire regarding sensation, nipple satisfaction, and breast symptoms
Post-operative-two-year Quality of life | Two-year after breast reconstructive surgery
  Patient-reported outcome assessed by the BREAST-Q™ Reconstruction module questionnaire and a additional questionnaire regarding sensation, nipple satisfaction, and breast symptoms
Post-operative-one-year Quality of life | One-year after breast reconstructive surgery
  Patient-reported outcome assessed by the BREAST-Q™ Reconstruction module questionnaire and a additional questionnaire regarding sensation, nipple satisfaction, and breast symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Patient privacy